CLINICAL TRIAL: NCT03140449
Title: Study of Combination Therapy With Topical Rapamycin and Calcitriol for Cutaneous Lesions of Tuberous Sclerosis: A Double-blind Randomized Controlled Trial
Brief Title: Topical Rapamycin and Calcitriol for Angiofibroma of Tuberous Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201306009MINB
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2013-09

CONDITIONS: Facial Angiofibroma
Keywords: Tuberous sclerosis complex; facial angiofibroma; rapamycin; calcitriol
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Sirolimus; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Rapamycin (Experimental): Rapamycin(0.1%)
  Interventions: Drug: Rapamycin
- Calcitriol (Experimental): Calcitriol(3mcg/g)
  Interventions: Drug: Calcitriol
- Rapamycin-calcitriol combination (Experimental): Rapamycin(0.1%) with Calcitriol(3mcg/g)
  Interventions: Drug: Rapamycin-calcitriol combination

INTERVENTIONS:
Drug: Rapamycin — topical rapamycin (0.1%) or calcitriol (3 mcg/g) single-agent therapy versus their combination were applied twice a day by a left-right randomized, split-face comparison for 12 weeks.
  In period 2, the patients entered an open-label study and were reassigned to use the more effective ointment on both cheeks for another 12 weeks (week 13-24).
  Other Names: Sirolimus
  Arms: Rapamycin
Drug: Calcitriol — topical rapamycin (0.1%) or calcitriol (3 mcg/g) single-agent therapy versus their combination were applied twice a day by a left-right randomized, split-face comparison for 12 weeks.
  In period 2, the patients entered an open-label study and were reassigned to use the more effective ointment on both cheeks for another 12 weeks (week 13-24).
  Other Names: Rocaltrol
  Arms: Calcitriol
Drug: Rapamycin-calcitriol combination — topical rapamycin (0.1%) or calcitriol (3 mcg/g) single-agent therapy versus their combination were applied twice a day by a left-right randomized, split-face comparison for 12 weeks.
  In period 2, the patients entered an open-label study and were reassigned to use the more effective ointment on both cheeks for another 12 weeks (week 13-24).
  Other Names: Sirolimus-Rocaltrol combination
  Arms: Rapamycin-calcitriol combination

SUMMARY:
The aim of the study is to determine the effect and safety of topical rapamycin or calcitriol and their combination for the treatment of TSC-associated facial angiofibroma.

Methods: A total of 52 TSC patients including 20 male and 32 female subjects were recruited, and 50 of them completed the period 1 study. In period 1, topical rapamycin (0.1%) or calcitriol (3 mcg/g) single-agent therapy versus their combination were applied twice a day by a left-right randomized, split-face comparison for 12 weeks. The primary end point was the reduction of facial angiofibroma severity index (FASI) for the grade of erythema, papule size, elevation and extension of the lesions at week 12. In period 2, the patients entered an open-label study and were reassigned to use the more effective ointment on both cheeks for another 12 weeks (week 13-24). A follow-up FASI analysis for recurrence after drug discontinuance for 12 weeks was also performed (week 36). The secondary end point was the reduction of Visual Analysis Score (VAS) evaluated by the subjects themselves at week 12.

DETAILED DESCRIPTION:
Background: Tuberous sclerosis complex (TSC)-associated facial angiofibroma is psychologically debilitating to both patients and their family members. The pathogenesis of TSC stems from TSC1 or TSC2 mutations, leading to the defect in mechanistic target of rapamycin (mTOR) inhibition. Rapamycin is an mTOR inhibitor and is effective for TSC facial angiofibroma through topical administration. Calcitriol, a vitamin D3 analogue, has been shown to lessen skin fibrosis in scleroderma and may be therapeutically beneficial to angiofibromas.

Objectives: The aim of the study is to determine the effect and safety of topical rapamycin or calcitriol and their combination for the treatment of TSC-associated facial angiofibroma.

Methods: A total of 52 TSC patients including 20 male and 32 female subjects were recruited, and 50 of them completed the period 1 study. In period 1, topical rapamycin (0.1%) or calcitriol (3 mcg/g) single-agent therapy versus their combination were applied twice a day by a left-right randomized, split-face comparison for 12 weeks. The primary end point was the reduction of facial angiofibroma severity index (FASI) for the grade of erythema, papule size, elevation and extension of the lesions at week 12. In period 2, the patients entered an open-label study and were reassigned to use the more effective ointment on both cheeks for another 12 weeks (week 13-24). A follow-up FASI analysis for recurrence after drug discontinuance for 12 weeks was also performed (week 36). The secondary end point was the reduction of Visual Analysis Score (VAS) evaluated by the subjects themselves at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have been diagnosed or highly suspected as having TSC.
2. Subjects must be aged 7 to 70 years at Screening, and can be either sex.
3. Subjects must have symmetric facial angiofibromas.

Exclusion Criteria:

1. Pregnancy or with a plan to be pregnant.
2. Subjects who cannot comply the treatment protocol.
3. Subjects with kidney or liver/ biliary dysfunction.
4. Subjects with hypercalcaemia and patients known to suffer from abnormal calcium metabolism.
5. Subjects on systemic treatment of calcium deficiency.
6. Subjects known to be hypersensitive to rapamycin or calcitriol.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
facial angioﬁbroma severity index (FASI) | at week 12
  the reduction of facial angioﬁbroma severity index (FASI) for the grade of erythema, papule size, elevation and extension of the lesions at week 12

CONTACTS AND LOCATIONS:
Overall Officials: YI-HUA LIAO, A.P., Principal Investigator — A.P.

IPD SHARING:
Plan to Share IPD: Undecided